CLINICAL TRIAL: NCT04060823
Title: Implementing a Healthcare Provider Education Intervention in Rural Communities to Reduce Asthma Morbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201803077
Record Dates: First submitted 2019-08-16; First posted 2019-08-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Easy Breathing (Experimental): Easy Breathing will be implemented in participating clinics. Asthma-related sick visits will be monitored for changes.
  Interventions: Other: Easy Breathing program

INTERVENTIONS:
Other: Easy Breathing program — Easy Breathing is a longstanding, nationally recognized program that translates asthma management guidelines into a standardized and usable format for healthcare providers. As part of the program primary healthcare providers will identify children at-risk for adverse asthma outcomes and provide care coordination services. Patients receive a tailored, comprehensive Asthma Treatment Plan with information regarding daily medication use and management of acute symptoms based on asthma severity.

SUMMARY:
The aim of the study is to pilot test the implementation of healthcare provider education interventions to improve asthma outcomes in rural youth residing in Bradford County, Florida. The investigators propose to assess the feasibility and acceptability of implementing the Easy Breathing program a rural, medically underserved county and evaluate changes in healthcare provider practices and asthma-related outcomes of rural youth diagnosed with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Any child between 6 months and 18 years of age at one of the primary care clinics in Braford county.

Exclusion Criteria:

* Unable to meet inclusion criteria.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 512 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in child asthma diagnosis rates | Baseline up to Year 1
  Asthma diagnosis yearly rates (number of children newly diagnosed / number of children seen per year) will be compared before and after implementation of the Easy Breathing program.

CONTACTS AND LOCATIONS:
Overall Officials: David A Fedele, PhD, Principal Investigator — University of Florida
Locations (4):
- United States (4):
  - Bradford County Health Department, Starke, Florida
  - Shands Starke Medical Group, Starke, Florida
  - Southside Elementary School, Starke, Florida
  - Starke Elementary School, Starke, Florida

IPD SHARING:
Plan to Share IPD: No